CLINICAL TRIAL: NCT01051661
Title: A Study to Evaluate the Safety and Efficacy of A/California/7/2009 (H1N1)V-like Vaccines GSK2340274A and GSK2340273A in Children Aged 6 Months to Less Than 10 Years of Age
Brief Title: Safety and Efficacy of H1N1 Vaccines in Children Aged 6 Months to Less Than 10 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 114000
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Influenza
Keywords: Influenza; H1N1; Pandemic
MeSH Terms: conditions — Influenza, Human | interventions — arepanrix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Arepanrix 2D 6M-3Y Group (Experimental): Subjects, male and female, aged 6 months (M) to 3 years (Y), received 2 doses (D) of the Arepanrix™ vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340274A (alternative formulations)
- Arepanrix 2D 3Y-10Y Group (Experimental): Subjects, male and female, aged 3 years (Y) to 10 years, received 2 doses (D) of the Arepanrix™ vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340274A (alternative formulations)
- Arepanrix 1D 6M-3Y Group (Experimental): Subjects, male and female, aged 6 months (M) to 3 years (Y), received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340274A (alternative formulations); Biological: Placebo
- Arepanrix 1D 3Y-10Y Group (Experimental): Subjects, male and female, aged 3 years (Y) to 10 years, received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340274A (alternative formulations); Biological: Placebo
- GSK2340273A 6M-3Y Group (Experimental): Subjects, male and female, aged 6 months (M) to 3 years (Y), received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340273A (alternative formulations)
- GSK2340273A 3Y-10Y Group (Experimental): Subjects, male and female, aged 3 years (Y) to 10 years, received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340273A (alternative formulations)

INTERVENTIONS:
Biological: GSK Biologicals' investigational vaccine GSK2340274A (alternative formulations) — Intramuscular injection, one or two doses
  Other Names: Arepanrix
  Arms: Arepanrix 1D 3Y-10Y Group; Arepanrix 1D 6M-3Y Group; Arepanrix 2D 3Y-10Y Group; Arepanrix 2D 6M-3Y Group
Biological: GSK Biologicals' investigational vaccine GSK2340273A (alternative formulations) — Intramuscular injection, two doses
  Arms: GSK2340273A 3Y-10Y Group; GSK2340273A 6M-3Y Group
Biological: Placebo — Intramuscular injection, one dose
  Arms: Arepanrix 1D 3Y-10Y Group; Arepanrix 1D 6M-3Y Group

SUMMARY:
The purpose of this study is to characterize the safety and efficacy of GSK Biologicals' H1N1 flu candidate vaccines GSK2340274A and GSK2340273A in children 6 months to less than 10 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children 6 months to less than 10 years of age at the time of the first vaccination. "Less than 10 years of age" implies inclusion of children who have not reached their 10th birthday as of Day 0, the day of first vaccine dose under this protocol.
* Written informed consent obtained from the subject's parent(s)/legally acceptable representative(s) (LAR(s)); written informed assent obtained from the subject if appropriate pre local requirements).
* Stable health status as defined by absence of a health event satisfying the definition of a SAE, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within 1 month prior to enrolment.
* Parent(s)/LAR(s) available and accessible for active surveillance contacts.
* Parent(s)/LAR(s) and (if age-appropriate, subjects) who, in the investigator's opinion, can and will comply with the requirements of the protocol as documented by signature on the informed consent document.
* Female subjects of non-childbearing potential (pre-menarche) may be enrolled in the study.

Exclusion Criteria:

* Previous vaccination with an A/California/7/2009 (H1N1)v-like virus vaccine.
* Medical history of physician-confirmed infection with an A/California/7/2009 (H1N1)v-like virus.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject or parent(s)/LAR(s) unable/unlikely to provide accurate safety reports.
* Presence of a temperature ≥ 38.0ºC (≥ 100.4ºF) by any route or method, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment (first dose of study vaccine), or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articular or inhaled glucocorticoids are allowed.
* Receipt of any immunoglobulins and/or any blood products within 6 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin are eligible if no such doses are given in the 24 hours before a study vaccination. Persons receiving prophylactic antiplatelet medications, e.g., low-dose acetylsalicylic acid, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Administration of any licensed live attenuated vaccine within 4 weeks before the first vaccination or of any licensed inactivated vaccine within 2 weeks before the first vaccination.
* Planned administration of any vaccine not foreseen by the study protocol between Day 0 and Day 42. Routine childhood vaccinations are exempted if they cannot be delayed, but they must not be administered on the same day as the H1N1 vaccine candidate.
* Planned use of a pandemic monovalent A/California/7/2009 (H1N1)v-like virus vaccine other than the study vaccines during the study period.
* Planned administration of seasonal trivalent influenza vaccine during the 4 month period following Day 0.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days before the first dose of study vaccine, or planned use during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines (including egg proteins or mercurial preservatives); a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Child in care.

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6154 (Actual)
Dates: Start 2010-02-12 (Actual); Primary Completion 2011-08-31 (Actual); Study Completion 2011-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Australia (2):
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Carlton, Victoria
- Brazil (2):
  - GSK Investigational Site, Florianópolis, Santa Catarina
  - GSK Investigational Site, São Paulo
- GSK Investigational Site, Cali, Colombia
- GSK Investigational Site, San José, Costa Rica
- Mexico (4):
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Monterrey
- Philippines (3):
  - GSK Investigational Site, City of Muntinlupa
  - GSK Investigational Site, Dasmariñas, Cavite
  - GSK Investigational Site, Sampaloc, Manila
- GSK Investigational Site, Singapore, Singapore
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Nolan T, Roy-Ghanta S, Montellano M, Weckx L, Ulloa-Gutierrez R, Lazcano-Ponce E, Kerdpanich A, Safadi MA, Cruz-Valdez A, Litao S, Lim FS, de Los Santos AM, Weber MA, Tinoco JC, Mezerville MH, Faingezicht I, Kosuwon P, Lopez P, Borja-Tabora C, Li P, Durviaux S, Fries L, Dubin G, Breuer T, Innis BL, Vaughn DW. Relative efficacy of AS03-adjuvanted pandemic influenza A(H1N1) vaccine in children: results of a controlled, randomized efficacy trial. J Infect Dis. 2014 Aug 15;210(4):545-57. doi: 10.1093/infdis/jiu173. Epub 2014 Mar 20. PMID 24652494
- [Derived] Taylor S, Lopez P, Weckx L, Borja-Tabora C, Ulloa-Gutierrez R, Lazcano-Ponce E, Kerdpanich A, Angel Rodriguez Weber M, Mascarenas de Los Santos A, Tinoco JC, Safadi MA, Lim FS, Hernandez-de Mezerville M, Faingezicht I, Cruz-Valdez A, Feng Y, Li P, Durviaux S, Haars G, Roy-Ghanta S, Vaughn DW, Nolan T. Respiratory viruses and influenza-like illness: Epidemiology and outcomes in children aged 6 months to 10 years in a multi-country population sample. J Infect. 2017 Jan;74(1):29-41. doi: 10.1016/j.jinf.2016.09.003. Epub 2016 Sep 22. PMID 27667752
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114000 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114000 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114000 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114000 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114000 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114000 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 1654 subjects enrolled, study vaccine was not administered but subject number was allocated to 9 subjects. These 9 subjects were excluded from the study, therefore leading to 1645 subjects starting the study.
Period: Overall Study
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Started | 610 | 1438 | 612 | 1436 | 613 | 1436
Completed | 576 | 1375 | 573 | 1380 | 578 | 1369
Not Completed | 34 | 63 | 39 | 56 | 35 | 67
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 13 | 22 | 15 | 17 | 10 | 24
Not completed — Migrated/moved from study area | 1 | 6 | 6 | 8 | 7 | 3
Not completed — Refused blood sampling | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Data not reliable | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Unable to attend visit(s) | 2 | 4 | 2 | 1 | 3 | 2
Not completed — Consent not received from both parents | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Failure to comply with protocol | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Subject lost legal representation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 16 | 30 | 13 | 28 | 12 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group | Total
Number analyzed (Participants) | 610 | 1438 | 612 | 1436 | 613 | 1436 | 6145
Age, Continuous [Mean (Standard Deviation); unit: Months] | 21.0 (8.8) | 73.4 (23.8) | 21.2 (8.8) | 73.2 (24.2) | 21.2 (8.6) | 73.2 (24.3) | 57.7 (31.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 291 | 688 | 308 | 748 | 291 | 732 | 3058
  Male | 319 | 750 | 304 | 688 | 322 | 704 | 3087
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage/African American | 8 | 22 | 4 | 22 | 3 | 26 | 85
  Asian-Central/South Asian Heritage | 0 | 1 | 1 | 0 | 0 | 2 | 4
  Asian-East Asian Heritage | 1 | 1 | 0 | 2 | 1 | 7 | 12
  Asian-Japanese Heritage | 1 | 2 | 0 | 3 | 0 | 2 | 8
  Asian-South East Asian Heritage | 297 | 507 | 301 | 503 | 297 | 499 | 2404
  Native Hawaiian or other Pacific islander | 0 | 2 | 1 | 0 | 0 | 1 | 4
  White-Arabic/North African Heritage | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White-Caucasian/European Heritage | 68 | 172 | 59 | 161 | 68 | 165 | 693
  Other | 235 | 731 | 246 | 745 | 243 | 734 | 2934

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting at Least One A/California Influenza Event
Description: The influenza virus presence was confirmed by quantitative reverse transcription polymerase chain reaction assay (RT-qPCR).
Time Frame: From 14 days after first vaccination until study conclusion on Day 385
Population: The analyses were performed on the According-to-Protocol (ATP) cohort for analysis of efficacy, which included all eligible subjects, who received the study vaccine/placebo according to their treatment assignment, and for whom efficacy data were available. The groups were pooled, based on the type of vaccine received and regardless the age strata.
Measure: Count of Participants; unit: Participants
Groups:
- Arepanrix 2D Group: Subjects, male and female, aged 6 months to 10 years, received 2 doses (D) of the Arepanrix™ vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh. This group pooled the subjects from the 6M-3Y and 3Y-10Y age strata.
- Arepanrix 1D Group: Subjects, male and female, aged 6 months to 10 years, received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh. This group pooled the subjects from the 6M-3Y and 3Y-10Y age strata.
- GSK2340273A Group: Subjects, male and female, aged 6 months to 10 years, received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh. This group pooled the subjects from the 6M-3Y and 3Y-10Y age strata.
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 3 | 7 | 13
Statistical Analysis 1: Comparison: Arepanrix 2D Group vs GSK2340273A Group; Evaluation of the relative protective efficacy of 2 doses of Arepanrix™ vaccine (Arepanrix 2D Group) compared to two doses of GSK2340273A vaccine (GSK2340273A Group) beginning 14 days after Dose 1 vaccination (for each subject enrolled) and continuing until study conclusion on Day 385; Test type: Superiority — The non-inferiority objective was met if the lower limit (LL) of the 95% CI for the Vaccine Efficacy Improvement (VEI) was > -33%. Furthermore, the superiority objective was met if the LL of the 95% CI for the VEI was >0; Vaccine efficacy increase = 76.70, 95% CI 2-sided [18.53 to 93.39]

2. Secondary Outcome: Number of Subjects Reporting at Least One A/California Influenza Event
Description: as for outcome 1
Time Frame: From 42 days after first vaccination until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 3 | 5 | 9

3. Secondary Outcome: Number of Subjects Reporting at Least One A/California Influenza Event
Description: as for outcome 1
Time Frame: From Day 0 until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 4 | 9 | 13

4. Secondary Outcome: Number of Subjects Reporting at Least One Culture Confirmed A/California Influenza Event
Description: The influenza virus presence was confirmed by a positive culture.
Time Frame: From 14 days after first vaccination until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 2 | 6 | 8

5. Secondary Outcome: Number of Subjects Reporting at Least One Culture Confirmed A/California Influenza Event
Description: The influenza virus presence was confirmed by a positive culture.
Time Frame: From 42 days after first vaccination until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 2 | 4 | 5

6. Secondary Outcome: Number of Subjects Reporting at Least One Culture Confirmed A/California Influenza Event
Description: The influenza virus presence was confirmed by a positive culture.
Time Frame: From Day 0 until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 3 | 7 | 8

7. Secondary Outcome: Number of Subjects With at Least One Pneumonia Event
Time Frame: From 14 days after first vaccination until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 16 | 13 | 20

8. Secondary Outcome: Number of Subjects With at Least One Pneumonia Event
Time Frame: From 42 days after first vaccination until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 16 | 12 | 18

9. Secondary Outcome: Number of Subjects With at Least One Pneumonia Event
Time Frame: From Day 0 after first vaccination until study conclusion on Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 16 | 15 | 22

10. Secondary Outcome: Number of Subjects With at Least One Pneumonia Event
Description: Pneumonia was confirmed by quantitative reverse transcription polymerase chain reaction assay (RT-qPCR).
Time Frame: From 14 days after first vaccination until study conclusion at Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 0 | 0 | 0

11. Secondary Outcome: Number of Subjects With at Least One Pneumonia Event
Description: Pneumonia was confirmed by quantitative reverse transcription polymerase chain reaction assay (RT-qPCR).
Time Frame: From 42 days after first vaccination until study conclusion at Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 0 | 0 | 0

12. Secondary Outcome: Number of Subjects With at Least One Pneumonia Event
Description: Pneumonia was confirmed by quantitative reverse transcription polymerase chain reaction assay (RT-qPCR).
Time Frame: From Day 0 after first vaccination until study conclusion at Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1940 | 1933 | 1930
Participants | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With Protocol Specified Influenza-like Illness (ILI) Symptoms in All Reported ILI Cases
Description: Protocol specified ILI symptoms were: fever, muscle aches all over the body, cough, sore throat, runny or stuffy nose, short of breath, headache, vomiting, diarrhea, chills and fatigue.
Time Frame: From Day 0 until study end at Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1903 | 1913 | 1897
Participants
  Fever | 745 | 685 | 700
  Muscle aches all over body | 271 | 219 | 239
  Cough | 668 | 626 | 634
  Sore throat | 395 | 362 | 379
  Runny or stuffy nose | 682 | 628 | 649
  Short of breath | 236 | 227 | 352
  Headache | 360 | 340 | 422
  Vomiting | 311 | 265 | 301
  Diarrhea | 132 | 141 | 160
  Chills | 282 | 265 | 272
  Fatigue | 347 | 314 | 326

14. Secondary Outcome: Number of Subjects With Protocol Specified Influenza-like Illness (ILI) Symptoms in All Reported ILI Cases
Description: Protocol specified ILI symptoms were: fever, muscle aches all over the body, cough, sore throat, runny or stuffy nose, short of breath, headache, vomiting, diarrhea, chills and fatigue. Analysis for the time frame Day 42 till Day 385 was not performed as planned per protocol.
Time Frame: From Day 14 until study end at Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1903 | 1913 | 1897
Participants
  Fever | 716 | 659 | 677
  Muscle aches all over body | 264 | 210 | 227
  Cough | 643 | 599 | 614
  Sore throat | 382 | 351 | 360
  Runny or stuffy nose | 656 | 605 | 627
  Short of breath | 225 | 218 | 214
  Headache | 348 | 329 | 344
  Vomiting | 302 | 254 | 291
  Diarrhea | 124 | 137 | 157
  Chills | 278 | 255 | 266
  Fatigue | 340 | 302 | 314

15. Secondary Outcome: Number of Subjects With Protocol Specified ILI Symptoms in RT-qPCR-confirmed A/California Influenza Cases
Description: as for outcome 13
Time Frame: From Day 0 until study end at Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1903 | 1913 | 1897
Participants
  Fever | 4 | 7 | 11
  Muscle aches all over body | 0 | 2 | 4
  Cough | 4 | 7 | 11
  Sore throat | 1 | 3 | 6
  Runny or stuffy nose | 4 | 7 | 10
  Short of breath | 1 | 1 | 2
  Headache | 0 | 5 | 7
  Vomiting | 2 | 2 | 4
  Diarrhea | 1 | 3 | 2
  Chills | 2 | 3 | 5
  Fatigue | 2 | 4 | 4

16. Secondary Outcome: Number of Subjects With Protocol Specified ILI Symptoms in RT-qPCR-confirmed A/California Influenza Cases
Description: as for outcome 14
Time Frame: From Day 14 until study end at Day 385
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 1903 | 1913 | 1897
Participants
  Fever | 3 | 6 | 11
  Muscle aches all over body | 0 | 2 | 4
  Cough | 3 | 6 | 11
  Sore throat | 0 | 3 | 6
  Runny or stuffy nose | 3 | 6 | 10
  Short of breath | 1 | 1 | 2
  Headache | 0 | 4 | 7
  Vomiting | 2 | 2 | 4
  Diarrhea | 1 | 3 | 2
  Chills | 2 | 3 | 5
  Fatigue | 2 | 3 | 4

17. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day follow-up period (Day 0 - Day 6) after each dose and across doses
Population: The analyses were performed on the Total Vaccinated cohort, which included all subjects, from the age strata groups, who received at least 1 dose of study vaccine and who filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Groups:
- Arepanrix 2D 6M-3Y Group: Subjects, male and female, aged 6 months (M) to less than (<) 3 years (Y), received 2 doses (D) of the Arepanrix™ vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh.
- Arepanrix 2D 3Y-6Y Group: Subjects, male and female, aged 3 years (Y) to less than (<) 6 years, received 2 doses (D) of the Arepanrix™ vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
- Arepanrix 2D 6Y-10Y Group: Subjects, male and female, aged 6 years (Y) to less than (<) 10 years, received 2 doses (D) of the Arepanrix™ vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
- Arepanrix 1D 6M-3Y Group: Subjects, male and female, aged 6 months (M) to less than (<) 3 years (Y), received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh.
- Arepanrix 1D 3Y-6Y Group: Subjects, male and female, aged 3 years (Y) to less than (<) 6 years, received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
- Arepanrix 1D 6Y-10Y Group: Subjects, male and female, aged 6 years (Y) to less than (<) 10 years, received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
- GSK2340273A 6M-3Y Group: Subjects, male and female, aged 6 months (M) to less than (<) 3 years (Y), received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh.
- GSK2340273A 3Y-6Y Group: Subjects, male and female, aged 2 years (Y) to less than (<) 6 years, received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
- GSK2340273A 6Y-10Y Group: Subjects, male and female, aged 6 years (Y) to less than (<) 10 years, received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-6Y Group | Arepanrix 2D 6Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-6Y Group | Arepanrix 1D 6Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-6Y Group | GSK2340273A 6Y-10Y Group
Number analyzed (Participants) | 610 | 726 | 712 | 612 | 744 | 692 | 613 | 714 | 722
Participants
  Any Pain, Dose 1 | 204 | 369 | 416 | 189 | 357 | 409 | 122 | 212 | 254
  Grade 3 Pain, Dose 1 | 13 | 16 | 16 | 13 | 24 | 25 | 5 | 7 | 6
  Any Redness, Dose 1 | 8 | 9 | 13 | 8 | 8 | 18 | 1 | 2 | 4
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any Swelling, Dose 1 | 11 | 30 | 25 | 17 | 16 | 30 | 2 | 10 | 13
  Grade 3 Swelling, Dose 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 592 | 708 | 699 | 591 | 727 | 681 | 593 | 696 | 709
  Any Pain, Dose 2 | 213 | 344 | 347 | 104 | 153 | 133 | 86 | 157 | 213
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 592 | 708 | 699 | 591 | 727 | 681 | 593 | 696 | 709
  Grade 3 Pain, Dose 2 | 14 | 24 | 23 | 5 | 5 | 5 | 5 | 6 | 5
  Any Redness, Dose 2: number analyzed (Participants) | 592 | 708 | 699 | 591 | 727 | 681 | 593 | 696 | 709
  Any Redness, Dose 2 | 12 | 7 | 17 | 1 | 1 | 1 | 1 | 0 | 3
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 592 | 708 | 699 | 591 | 727 | 681 | 593 | 696 | 709
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 592 | 708 | 699 | 591 | 727 | 681 | 593 | 696 | 709
  Any Swelling, Dose 2 | 24 | 19 | 21 | 1 | 4 | 4 | 2 | 8 | 7
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 592 | 708 | 699 | 591 | 727 | 681 | 593 | 696 | 709
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 288 | 454 | 487 | 222 | 382 | 431 | 154 | 258 | 322
  Grade 3 Pain, Across doses | 24 | 39 | 34 | 16 | 28 | 27 | 10 | 11 | 10
  Any Redness, Across doses | 20 | 16 | 25 | 8 | 8 | 18 | 2 | 2 | 6
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Any Swelling, Across doses | 31 | 42 | 38 | 17 | 17 | 32 | 3 | 16 | 15
  Grade 3 Swelling, Across doses | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

18. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms in Children Aged 6 Months to Less Than 6 Years
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and temperature [defined as axillary temperature equal to or above (≥) 38.0 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness which prevented normal everyday activity. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 temperature = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day follow-up period (Day 0 - Day 6) after each dose and across doses
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-6Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-6Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-6Y Group
Number analyzed (Participants) | 610 | 726 | 612 | 744 | 613 | 714
Participants
  Any Drowsiness, Dose 1 | 105 | 103 | 93 | 112 | 106 | 101
  Grade 3 Drowsiness, Dose 1 | 7 | 7 | 3 | 1 | 3 | 5
  Related Drowsiness, Dose 1 | 62 | 70 | 50 | 74 | 56 | 62
  Any Irritability, Dose 1 | 149 | 99 | 128 | 111 | 135 | 67
  Grade 3 Irritability, Dose 1 | 5 | 3 | 3 | 1 | 2 | 1
  Related Irritability, Dose 1 | 97 | 70 | 82 | 80 | 83 | 43
  Any Loss of appetite, Dose 1 | 109 | 106 | 89 | 97 | 116 | 82
  Grade 3 Loss of appetite, Dose 1 | 7 | 5 | 5 | 4 | 8 | 5
  Related Loss of appetite, Dose 1 | 68 | 64 | 51 | 63 | 63 | 45
  Any Temperature, Dose 1 | 77 | 59 | 88 | 55 | 45 | 33
  Grade 3 Temperature, Dose 1 | 18 | 7 | 21 | 15 | 18 | 3
  Related Temperature, Dose 1 | 45 | 40 | 63 | 39 | 25 | 16
  Any Drowsiness, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Any Drowsiness, Dose 2 | 115 | 92 | 53 | 58 | 73 | 59
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Grade 3 Drowsiness, Dose 2 | 8 | 3 | 3 | 3 | 6 | 1
  Related Drowsiness, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Related Drowsiness, Dose 2 | 81 | 65 | 32 | 42 | 52 | 41
  Any Irritability, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Any Irritability, Dose 2 | 164 | 95 | 81 | 63 | 104 | 48
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Grade 3 Irritability, Dose 2 | 9 | 2 | 2 | 2 | 6 | 2
  Related Irritability, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Related Irritability, Dose 2 | 114 | 72 | 44 | 46 | 64 | 34
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Any Loss of appetite, Dose 2 | 112 | 96 | 61 | 67 | 102 | 53
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Grade 3 Loss of appetite, Dose 2 | 10 | 2 | 7 | 2 | 6 | 2
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Related Loss of appetite, Dose 2 | 73 | 56 | 27 | 49 | 62 | 34
  Any Temperature, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Any Temperature, Dose 2 | 148 | 99 | 44 | 47 | 56 | 31
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Grade 3 Temperature, Dose 2 | 29 | 11 | 12 | 10 | 14 | 4
  Related Temperature, Dose 2: number analyzed (Participants) | 592 | 708 | 591 | 727 | 593 | 696
  Related Temperature, Dose 2 | 113 | 74 | 22 | 27 | 28 | 19
  Any Drowsiness, Across doses | 175 | 160 | 124 | 137 | 149 | 133
  Grade 3 Drowsiness, Across doses | 15 | 10 | 6 | 4 | 8 | 6
  Related Drowsiness, Across doses | 120 | 116 | 71 | 97 | 92 | 89
  Any Irritability, Across doses | 237 | 160 | 164 | 139 | 190 | 95
  Grade 3 Irritability, Across doses | 14 | 5 | 5 | 3 | 8 | 2
  Related Irritability, Across doses | 163 | 120 | 104 | 109 | 121 | 66
  Any Loss of appetite, Across doses | 182 | 170 | 126 | 134 | 175 | 115
  Grade 3 Loss of appetite, Across doses | 16 | 7 | 12 | 6 | 14 | 7
  Related Loss of appetite, Across doses | 122 | 109 | 71 | 94 | 109 | 69
  Any Temperature, Across doses | 198 | 145 | 124 | 97 | 97 | 59
  Grade 3 Temperature, Across doses | 47 | 18 | 33 | 25 | 30 | 6
  Related Temperature, Across doses | 143 | 107 | 83 | 62 | 51 | 34

19. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms in Children Aged Between 6 to 10 Years
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (gastro.sympt.), headache, joint pain at other location, muscle aches, shivering, sweating and temperature [defined as axillary temperature equal to or above (≥) 38.0 degrees Celsius (°C)]. Any = Incidence of a particular symptom regardless of intensity grade or relationship to study vaccination. Grade 3 = symptom which prevented normal everyday activity. Grade 3 temperature = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day follow-up period (Day 0 - Day 6) after each dose and across doses
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Groups:
- Arepanrix 2D 6Y-10Y Group: Subjects, male and female, aged 6 years (Y) to 10 years, received 2 doses (D) of the Arepanrix™ vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
- Arepanrix 1D 6Y-10Y Group: Subjects, male and female, aged 6 years (Y) to 10 years, received 1 dose (D) of the Arepanrix™ vaccine followed by 1 dose of saline placebo at a 21-day interval at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
- GSK2340273A 6Y-10Y Group: Subjects, male and female, aged 6 years (Y) to 10 years, received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
Arm/Group | Arepanrix 2D 6Y-10Y Group | Arepanrix 1D 6Y-10Y Group | GSK2340273A 6Y-10Y Group
Number analyzed (Participants) | 712 | 692 | 722
Participants
  Any Fatigue, Dose 1 | 90 | 82 | 81
  Grade 3 Fatigue, Dose 1 | 6 | 4 | 5
  Related Fatigue, Dose 1 | 65 | 52 | 42
  Any Gastro.sympt., Dose 1 | 41 | 45 | 49
  Grade 3 Gastro.sympt., Dose 1 | 5 | 2 | 4
  Related Gastro.sympt., Dose 1 | 22 | 27 | 15
  Any Headache, Dose 1 | 141 | 129 | 108
  Grade 3 Headache, Dose 1 | 9 | 3 | 5
  Related Headache, Dose 1 | 103 | 87 | 63
  Any Joint pain at other location, Dose 1 | 63 | 65 | 45
  Grade 3 Joint pain at other location, Dose 1 | 3 | 2 | 0
  Related Joint pain at other location, Dose 1 | 46 | 43 | 28
  Any Muscle aches, Dose 1 | 105 | 116 | 67
  Grade 3 Muscle aches, Dose 1 | 5 | 6 | 0
  Related Muscle aches, Dose 1 | 81 | 84 | 44
  Any Shivering, Dose 1 | 28 | 31 | 18
  Grade 3 Shivering, Dose 1 | 2 | 1 | 2
  Related Shivering, Dose 1 | 21 | 19 | 6
  Any Sweating, Dose 1 | 27 | 29 | 33
  Grade 3 Sweating, Dose 1 | 2 | 1 | 2
  Related Sweating, Dose 1 | 18 | 14 | 13
  Any Temperature, Dose 1 | 34 | 32 | 21
  Grade 3 Temperature, Dose 1 | 7 | 8 | 4
  Related Temperature, Dose 1 | 26 | 19 | 10
  Any Fatigue, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Fatigue, Dose 2 | 89 | 51 | 48
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Fatigue, Dose 2 | 10 | 1 | 2
  Related Fatigue, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Fatigue, Dose 2 | 68 | 37 | 26
  Any Gastro.sympt., Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Gastro.sympt., Dose 2 | 34 | 28 | 33
  Grade 3 Gastro.sympt., Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Gastro.sympt., Dose 2 | 2 | 3 | 2
  Related Gastro.sympt., Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Gastro.sympt., Dose 2 | 23 | 19 | 17
  Any Headache, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Headache, Dose 2 | 148 | 75 | 75
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Headache, Dose 2 | 9 | 3 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Headache, Dose 2 | 105 | 48 | 45
  Any Joint pain at other location, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Joint pain at other location, Dose 2 | 61 | 35 | 23
  Grade 3 Joint pain at other location, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Joint pain at other location, Dose 2 | 5 | 3 | 1
  Related Joint pain at other location, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Joint pain at other location, Dose 2 | 42 | 28 | 13
  Any Muscle aches, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Muscle aches, Dose 2 | 105 | 48 | 46
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Muscle aches, Dose 2 | 7 | 3 | 1
  Related Muscle aches, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Muscle aches, Dose 2 | 82 | 41 | 35
  Any Shivering, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Shivering, Dose 2 | 34 | 15 | 10
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Shivering, Dose 2 | 1 | 2 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Shivering, Dose 2 | 22 | 10 | 7
  Any Sweating, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Sweating, Dose 2 | 36 | 15 | 20
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Sweating, Dose 2 | 3 | 2 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Sweating, Dose 2 | 25 | 6 | 8
  Any Temperature, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Any Temperature, Dose 2 | 61 | 16 | 19
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Grade 3 Temperature, Dose 2 | 14 | 5 | 4
  Related Temperature, Dose 2: number analyzed (Participants) | 699 | 681 | 709
  Related Temperature, Dose 2 | 42 | 5 | 11
  Any Fatigue, Across doses | 139 | 118 | 106
  Grade 3 Fatigue, Across doses | 14 | 5 | 7
  Related Fatigue, Across doses | 104 | 77 | 57
  Any Gastro.sympt., Across doses | 66 | 65 | 72
  Grade 3 Gastro.sympt., Across doses | 7 | 5 | 6
  Related Gastro.sympt., Across doses | 42 | 41 | 28
  Any Headache, Across doses | 231 | 170 | 158
  Grade 3 Headache, Across doses | 16 | 6 | 6
  Related Headache, Across doses | 168 | 115 | 95
  Any Joint pain at other location, Across doses | 102 | 92 | 61
  Grade 3 Joint pain at other location, Across doses | 7 | 5 | 1
  Related Joint pain at other location, Across doses | 73 | 67 | 37
  Any Muscle aches, Across doses | 165 | 140 | 98
  Grade 3 Muscle aches, Across doses | 11 | 9 | 1
  Related Muscle aches, Across doses | 131 | 107 | 68
  Any Shivering, Across doses | 56 | 42 | 27
  Grade 3 Shivering, Across doses | 3 | 3 | 2
  Related Shivering, Across doses | 38 | 27 | 12
  Any Sweating, Across doses | 51 | 41 | 44
  Grade 3 Sweating, Across doses | 5 | 2 | 2
  Related Sweating, Across doses | 36 | 20 | 17
  Any Temperature, Across doses | 89 | 44 | 37
  Grade 3 Temperature, Across doses | 21 | 13 | 7
  Related Temperature, Across doses | 63 | 22 | 19

20. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: Up to Day 385
Population: The analyses were performed on the Total Vaccinated cohort, which included all subjects, who received at least 1 dose of study vaccine and who filled in their symptom sheets. This analysis compared the different treatment groups based on the type of vaccine received.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 2048 | 2048 | 2049
Participants | 0 | 2 | 3

21. Secondary Outcome: Number of Subjects With Any Medically-attended Adverse Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: Up to Day 385
Population: The analyses were performed on the Total Vaccinated cohort, which included all subjects, who received at least 1 dose of study vaccine and who filled in their symptom sheets. The groups were pooled, based on the type of vaccine received and regardless the age strata.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 2048 | 2048 | 2049
Participants | 1189 | 1173 | 1190

22. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 to Day 42
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 2048 | 2048 | 2049
Participants | 913 | 904 | 895

23. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to Day 385
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D Group | Arepanrix 1D Group | GSK2340273A Group
Number analyzed (Participants) | 2048 | 2048 | 2049
Participants | 76 | 66 | 68

24. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Days 0 and 42
Population: The analyses were performed on the According-to-protocol (ATP) cohort for immunogenicity - Day 42, which included all evaluable subjects with both doses of study vaccine/placebo administered per protocol treatment assignment and assay results for antibodies against A/California at the relevant timepoints were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 233 | 167 | 232 | 156 | 223 | 164
Titers
  Day 0: number analyzed (Participants) | 229 | 166 | 228 | 153 | 220 | 161
  Day 0 | 12.40 [10.21 to 15.06] | 16.92 [13.77 to 20.80] | 11.19 [9.32 to 13.43] | 14.17 [11.48 to 17.49] | 12.25 [9.97 to 15.07] | 14.76 [12.04 to 18.10]
  Day 42 | 1738.90 [1598.65 to 1891.44] | 1345.36 [1228.32 to 1473.55] | 258.02 [219.86 to 302.79] | 279.52 [229.58 to 340.31] | 188.89 [156.13 to 228.53] | 443.98 [367.03 to 537.04]

25. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: A seropositive subject was defined as a subject whose HI titers were greater than or equal to (≥) 1:10.
Time Frame: At Days 0 and 42
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 233 | 167 | 232 | 156 | 223 | 164
Participants
  Day 0: number analyzed (Participants) | 229 | 166 | 228 | 153 | 220 | 161
  Day 0 | 66 | 82 | 62 | 69 | 60 | 73
  Day 42 | 233 | 167 | 232 | 156 | 220 | 163

26. Secondary Outcome: Number of Seroconverted (SCR) Subjects for Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: Seroconversion was defined as: for initially seronegative subjects, antibody titer ≥ 1:40 after vaccination; and for initially seropositive subjects, antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer.
Time Frame: At Day 42
Population: The analyses were performed on the According-to-protocol (ATP) cohort for immunogenicity - Day 42, which included all evaluable subjects from Arepanrix age strata groups and subjects from main GSK2340273A Group, with study vaccine/placebo administered per protocol and assay results available at the relevant timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 229 | 166 | 228 | 153 | 220 | 161
Participants | 228 | 166 | 224 | 149 | 187 | 155

27. Secondary Outcome: Number of Seroprotected (SPR) Subjects Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Days 0 and 42
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 233 | 167 | 232 | 156 | 223 | 164
Participants
  Day 0: number analyzed (Participants) | 229 | 166 | 228 | 153 | 220 | 161
  Day 0 | 61 | 66 | 55 | 45 | 55 | 53
  Day 42 | 233 | 167 | 229 | 154 | 199 | 160

28. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post-vaccination compared to Day 0.
Time Frame: At Day 42
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 229 | 166 | 228 | 153 | 220 | 161
Fold change | 140.8 [116.6 to 170.0] | 79.9 [65.3 to 97.6] | 23.4 [21.2 to 25.7] | 20.3 [17.7 to 23.3] | 15.6 [13.5 to 18.0] | 29.9 [25.1 to 35.7]

29. Secondary Outcome: Geometric Mean Antibody Titer Ratio Adjusted for Baseline Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1)
Description: The geometric mean titer ratio (GMT ratio) was defined as the ratio of geometric mean of the post-vaccination reciprocal HI titer between groups. The analysis was not performed for Day 182 and Day 385 as planned per protocol.
Time Frame: At Day 42
Population: The analyses were performed on the According-to-protocol (ATP) cohort for immunogenicity - Day 42, which included all evaluable subjects with study vaccine/placebo administered per protocol and assay results available at the relevant timepoint. The groups were pooled, based on the type of vaccine received and regardless the age strata.
Measure: Number; unit: Adjusted GMT ratio
Arm/Group | Arepanrix 1D Group | Arepanrix 2D Group | GSK2340273A Group
Number analyzed (Participants) | 381 | 395 | 381
Adjusted GMT ratio | 278.9 | 1548.5 | 275.8
Statistical Analysis 1: Comparison: Arepanrix 2D Group vs GSK2340273A Group; Adjusted Geometric mean titer (GMT) ratios of Hemagglutination Inhibition (HI) antibody post vaccination between Arepanrix 2D Group and GSK2340273A Group for A/California influenza strain (Arepanrix 2D Group/GSK2340273A Group); Test type: Other; Adjusted GMT ratios = 5.61, 95% CI 2-sided [4.92 to 6.41]
Statistical Analysis 2: Comparison: Arepanrix 1D Group vs GSK2340273A Group; Adjusted Geometric mean titer (GMT) ratios of Hemagglutination Inhibition (HI) antibody post vaccination between Arepanrix 1D Group and GSK2340273A Group for A/California influenza strain (Arepanrix 1D Group/GSK2340273A Group); Test type: Other; Adjusted GMT ratios = 1.05, 95% CI 2-sided [0.93 to 1.19]

30. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1)
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Days 0 and 182
Population: The analyses were performed on the According-to-protocol (ATP) cohort for immunogenicity - Day 182, which included all evaluable subjects from Arepanrix age strata groups and subjects from main GSK2340273A Group, with study vaccine/placebo administered per protocol and assay results available at the relevant timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 186 | 378 | 177 | 389 | 184 | 379
Titers
  Day 0: number analyzed (Participants) | 70 | 40 | 75 | 51 | 61 | 49
  Day 0 | 12.62 [8.79 to 18.12] | 11.79 [7.90 to 17.60] | 9.77 [7.23 to 13.22] | 17.57 [12.16 to 25.40] | 14.22 [9.03 to 22.40] | 12.19 [8.43 to 17.63]
  Day 182 | 287.22 [246.77 to 334.29] | 238.25 [213.25 to 266.18] | 76.52 [61.99 to 94.46] | 108.59 [94.10 to 125.30] | 74.94 [59.09 to 95.05] | 145.06 [128.28 to 164.03]

31. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: A seropositive subject was defined as a subject whose HI titers were greater than or equal to (≥) 1:10.
Time Frame: At Days 0 and 182
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 186 | 378 | 177 | 389 | 184 | 379
Participants
  Day 0: number analyzed (Participants) | 70 | 40 | 75 | 51 | 61 | 49
  Day 0 | 20 | 15 | 17 | 29 | 17 | 18
  Day 182 | 186 | 378 | 177 | 384 | 174 | 377

32. Secondary Outcome: Number of Seroconverted (SCR) Subjects for Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: as for outcome 26
Time Frame: At Day 182
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 70 | 40 | 75 | 51 | 61 | 49
Participants | 66 | 38 | 54 | 33 | 32 | 34

33. Secondary Outcome: Number of Seroprotected (SPR) Subjects Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Days 0 and 182
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 186 | 378 | 177 | 389 | 184 | 379
Participants
  Day 0: number analyzed (Participants) | 70 | 40 | 75 | 51 | 61 | 49
  Day 0 | 19 | 10 | 16 | 17 | 17 | 14
  Day 182 | 184 | 374 | 120 | 288 | 117 | 337

34. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: The seroconversion factor (SCF) was defined as the fold increase in serum Hemagglutination Inhibition (HI) geometric mean titers (GMTs) post vaccination compared to Day 0.
Time Frame: At Day 182
Population: as for outcome 30
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 70 | 40 | 75 | 51 | 61 | 49
Fold change | 24.0 [18.5 to 31.1] | 18.4 [13.1 to 25.8] | 8.0 [6.8 to 9.3] | 6.1 [4.7 to 7.9] | 4.8 [3.7 to 6.3] | 8.5 [6.4 to 11.4]

35. Secondary Outcome: Titers for Serum Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Days 0 and 385
Population: The analyses were performed on the According-to-protocol (ATP) cohort for immunogenicity - Day 385, which included all evaluable subjects from Arepanrix age strata groups and subjects from main GSK2340273A Group, with study vaccine/placebo administered per protocol and assay results available at the relevant timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 173 | 349 | 163 | 339 | 158 | 344
Titers
  Day 0: number analyzed (Participants) | 62 | 33 | 51 | 32 | 55 | 34
  Day 0 | 9.62 [6.76 to 13.69] | 15.71 [9.76 to 25.27] | 9.93 [6.71 to 14.71] | 14.92 [8.99 to 24.74] | 10.13 [7.04 to 14.56] | 13.57 [8.50 to 21.66]
  Day 385 | 265.61 [228.92 to 308.18] | 189.44 [169.64 to 211.55] | 112.56 [91.27 to 138.81] | 103.57 [89.90 to 119.32] | 54.90 [42.15 to 71.50] | 92.33 [80.18 to 106.31]

36. Secondary Outcome: Number of Seropositive Subjects for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: A seropositive subject was defined as a subject whose HI titers was greater than or equal to (≥) 1:10.
Time Frame: At Days 0 and 385
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 173 | 349 | 163 | 339 | 158 | 344
Participants
  Day 0: number analyzed (Participants) | 62 | 33 | 51 | 32 | 55 | 34
  Day 0 | 12 | 16 | 11 | 14 | 14 | 14
  Day 385 | 173 | 349 | 163 | 334 | 142 | 333

37. Secondary Outcome: Number of Seroconverted (SCR) Subjects for Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: as for outcome 26
Time Frame: At Day 385
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 62 | 33 | 51 | 32 | 55 | 34
Participants | 58 | 30 | 35 | 17 | 18 | 18

38. Secondary Outcome: Number of Seroprotected (SPR) Subjects Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: A seroprotected subject was defined as a vaccinated subject with serum Hemagglutination Inhibition (HI) titer ≥ 1:40.
Time Frame: At Days 0 and 385
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 173 | 349 | 163 | 339 | 158 | 344
Participants
  Day 0: number analyzed (Participants) | 62 | 33 | 51 | 32 | 55 | 34
  Day 0 | 11 | 12 | 10 | 10 | 11 | 9
  Day 385 | 169 | 339 | 128 | 266 | 82 | 259

39. Secondary Outcome: Seroconversion Factor for Hemagglutination Inhibition (HI) Antibodies Against Flu A/CAL/7/09 (H1N1) Influenza Strain
Description: as for outcome 34
Time Frame: At Day 385
Population: as for outcome 35
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
Number analyzed (Participants) | 62 | 33 | 51 | 32 | 55 | 34
Fold change | 26.6 [20.0 to 35.3] | 13.7 [9.9 to 19.0] | 8.5 [6.5 to 11.0] | 6.3 [4.2 to 9.4] | 3.7 [2.8 to 4.7] | 6.1 [4.2 to 8.7]

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms during the 7-day post-vaccination period (Days 0-6), Unsolicited AEs during the 42-day post-vaccination (Days 0-41), SAEs during the entire study period (Day 0 - Day 385).
Groups:
- GSK2340273A 6M-3Y Group: Subjects, male and female, aged 6 months to 3 years, received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified) or, for children <12 months of age, in the left anterolateral thigh. Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm) or, for, children <12 months of age, in the right anterolateral thigh.
- GSK2340273A 3Y-10Y Group: Subjects, male and female, aged 3 years to 10 years, received 2 doses (D) of the GSK2340273A vaccine at a 21-day interval (Days 0 and 21). First doses were administered in the deltoid region of the non-dominant arm (or left arm if dominance is not yet identified). Second doses were administered at a 21-day interval in the deltoid region of the dominant arm (or right arm).
Arm/Group | Arepanrix 2D 6M-3Y Group | Arepanrix 2D 3Y-10Y Group | Arepanrix 1D 6M-3Y Group | Arepanrix 1D 3Y-10Y Group | GSK2340273A 6M-3Y Group | GSK2340273A 3Y-10Y Group
All-Cause Mortality (participants affected / at risk) | 1/610 | 1/1438 | 1/612 | 0/1436 | 0/613 | 0/1436
Serious Adverse Events (participants affected / at risk) | 35/610 | 41/1438 | 29/612 | 37/1436 | 33/613 | 35/1436
Other Adverse Events (participants affected / at risk) | 498/610 | 1116/1438 | 439/612 | 1047/1436 | 446/613 | 891/1436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arepanrix 2D 6M-3Y Group (N=610) | Arepanrix 2D 3Y-10Y Group (N=1438) | Arepanrix 1D 6M-3Y Group (N=612) | Arepanrix 1D 3Y-10Y Group (N=1436) | GSK2340273A 6M-3Y Group (N=613) | GSK2340273A 3Y-10Y Group (N=1436)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drowning (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Ascariasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 7 (8) | 3 (3) | 7 (7) | 4 (4) | 11 (11) | 6 (6)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 3 (3) | 7 (8) | 2 (2) | 10 (10) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Typhoid fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (3) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 2 (2) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal laceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sexual abuse (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subgaleal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arepanrix 2D 6M-3Y Group (N=610) | Arepanrix 2D 3Y-10Y Group (N=1438) | Arepanrix 1D 6M-3Y Group (N=612) | Arepanrix 1D 3Y-10Y Group (N=1436) | GSK2340273A 6M-3Y Group (N=613) | GSK2340273A 3Y-10Y Group (N=1436)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 103 (125) | 0 (0) | 92 (101) | 1 (2) | 61 (69)
Decreased appetite (Metabolism and nutrition disorders) | 182 (222) | 171 (204) | 127 (151) | 135 (165) | 176 (219) | 115 (136)
Fatigue (General disorders) | 0 (0) | 140 (180) | 0 (0) | 118 (133) | 0 (0) | 106 (129)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 68 (77) | 2 (2) | 66 (74) | 0 (0) | 73 (83)
Headache (Nervous system disorders) | 4 (4) | 254 (321) | 4 (4) | 188 (224) | 0 (0) | 172 (205)
Irritability (Psychiatric disorders) | 237 (313) | 162 (196) | 164 (209) | 141 (176) | 190 (240) | 95 (115)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 166 (211) | 0 (0) | 140 (164) | 0 (0) | 100 (115)
Pain (General disorders) | 288 (417) | 941 (1476) | 222 (294) | 813 (1052) | 154 (208) | 580 (836)
Pyrexia (General disorders) | 230 (272) | 256 (279) | 151 (166) | 168 (186) | 128 (136) | 125 (137)
Somnolence (Nervous system disorders) | 175 (220) | 160 (195) | 124 (146) | 139 (172) | 149 (179) | 134 (161)
Swelling (General disorders) | 31 (35) | 80 (95) | 17 (18) | 49 (54) | 3 (4) | 31 (38)
Cough (Respiratory, thoracic and mediastinal disorders) | 61 (67) | 88 (100) | 47 (53) | 91 (98) | 56 (60) | 102 (111)
Diarrohoea (Gastrointestinal disorders) | 33 (36) | 23 (23) | 24 (26) | 28 (28) | 28 (30) | 20 (20)
Nasopharyngitis (Infections and infestations) | 99 (110) | 112 (120) | 82 (90) | 115 (126) | 98 (109) | 99 (107)
Upper respiratory tract infection (Infections and infestations) | 120 (135) | 132 (148) | 119 (129) | 144 (156) | 125 (147) | 127 (145)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.